CLINICAL TRIAL: NCT01783795
Title: Screening for Dent Disease Mutations in Patients With Proteinuria
Brief Title: Dent Disease Mutation Genotyping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Lieske, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10-006442; U54DK083908 (NIH)
Record Dates: First submitted 2013-01-23; First posted 2013-02-05 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Dent Disease
Keywords: Dent; Dents; Dent Disease; Dent genetic testing; CLCN5; OCRL1; Genetic testing for Dent Disease; Hereditary study for Dent Disease
MeSH Terms: conditions — Dent Disease | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetic Analysis (Other): Genetic Analysis
  Interventions: Other: Genetic Analysis

INTERVENTIONS:
Other: Genetic Analysis

SUMMARY:
This study will help the investigator determine whether certain genetic mutations, more than others, are a cause of more severe disease in Dent Disease.

DETAILED DESCRIPTION:
During this study visit, the investigator will draw one tube, about two teaspoonfuls (1 to 1 ½ teaspoons for children), of blood from the subject's arm to obtain white blood cells. These white blood cells will be used as a source of DNA for genetic testing. The investigator will use the isolated DNA to try to identify the gene that is defective in Dent Disease by comparing it with the structure of genes in normal individuals, patients with Dent Disease, and family members for Dent Disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed, or in the process of being diagnosed with Dent Disease.
* The patient has a family member diagnosed with Dent Disease.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with genetic mutations in either the CLCN5 or ORCL1 gene | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: John C. Lieske, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rare Kidney Stone Consortium — http://www.rarekidneystones.org